CLINICAL TRIAL: NCT04674150
Title: A Pilot Randomized Controlled Trial to Determine the Feasibility of Administering an auGmented reAlity gaMe to pediatrIc caNcer Patients underGoing Surgery (A GAMING Study)
Brief Title: A Pilot Randomized Controlled Trial for Feasibility of Administering an AR Game to Postoperative Pediatric Cancer Patients
Acronym: GAMING
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ALTality, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); M.D. Anderson Cancer Center (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARISE GAMING (Phase I); 1R42DA050365-01A1 (NIH)
Record Dates: First submitted 2020-12-08; First posted 2020-12-19 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Pediatric Cancer; Surgery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-AR Group (Sham Comparator): Patients allocated to the control group will be able to interact with the iPad and visualize objects and decals in the walls but not able to initiate the AR technology. In other terms, patients in this group will be provided with the same iPad to the AR group patients with the only exception that the AR technology will be off and will only see objects through the device camera in normal reality.
  Interventions: Device: ARISE without AR
- AR Group (Active Comparator): Patients randomized to the AR group will be able to use the iPad and SpellBound app to initiate the AR experiences in the game.
  Interventions: Device: ARISE with AR

INTERVENTIONS:
Device: ARISE with AR — An augmented reality game for mobile devices with AR experiences enabled
  Arms: AR Group
Device: ARISE without AR — An augmented reality game for mobile devices with AR experiences disabled as an control
  Arms: Non-AR Group

SUMMARY:
This is a pilot study to evaluate the feasibility of SpellBound's AR (augmented reality)-enabled scavenger hunt use among 20 pediatric cancer patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 3-18
2. English speaking parents/legal guardians and patients
3. Undergoing major surgery for cancer requiring postoperative hospitalization defined as ≥2 hours of duration of surgery and requiring postoperative hospital admission of at least one night
4. Expected to be prescribed postoperative inpatient opioids
5. Have never taken opioids or have had no daily opioid use within the last 30 days
6. Sufficient cognitive capacity to comprehend and interact with the game. This is defined as ability to utilize mobile technology (use iPad with or without assistance) and activate and respond to AR experiences within the app as determined by the clinician.
7. Both child and a legal guardian are willing and able to provide informed consent.

Exclusion Criteria:

1. History of documented peripheral neuropathy secondary to cancer treatment
2. Inability to demonstrate an understanding of the game from English instructions
3. Have previous played the ARISETM digital scavenger hunt game
4. Any additional concerns based on the study physicians' assessments

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who receive the AR game who are able to initiate the game and activate any targets with 1% error rate | The patient's postoperative inpatient hospital stay, average 7 days
  Success defined as at least 80% of patients who receive the AR game being able to initiate the game and activate any targets with 1% error rate

SECONDARY OUTCOMES:
Inpatient opioid use | The patient's postoperative inpatient hospital stay, average 7 days
  The average daily inpatient MEDD (morphine equivalent dose) will be calculated from the electronic medical record as previously used in pediatric cancer surgical patients by the investigator
Outpatient opioid use | The patient's postoperative inpatient hospital stay, average 7 days
  We will record whether the patient has any active opioid prescription 90-days (±10 Days) after surgery. This data will be confirmed by direct contact to patients' caregivers or via pharmacy registries on filled prescriptions.
Average daily inpatient pain score | The patient's postoperative inpatient hospital stay, average 7 days
  Age-appropriate pain-intensity scores will be determined using Visual and Colored Analogue Scales (VAS). This is a 10-point colored scaled validated for measuring pain intensity in pediatric populations and will be assessed twice daily at 9AM and 5PM.
Number of opioid requests (rescue analgesia) | The patient's postoperative inpatient hospital stay, average 7 days
  We will record the total number of times opioids were required by patients to nurses and the patient-controlled analgesia infusion pumps during the inpatient period as recorded in the electronic medical record.
Quality of life assessment | The patient's postoperative inpatient hospital stay, average 7 days
  Age-appropriate Pediatric Quality of Life Inventory (PedsQL) paper surveys will be administered to the patient (self-report) or guardian (proxy) when patients reach discharge-ready status.
Ambulation/ "out of bed" movement | The patient's postoperative inpatient hospital stay, average 7 days
  Distance (meters) achieved "out of bed" (ambulatory or non-ambulatory/wheelchair) during their inpatient stay while interacting with the app will be calculated by hand, based on how many times patient activated specific targets.
Discharge-ready status | The patient's postoperative inpatient hospital stay, average 7 days
  The number of days to discharge-ready status will be determined by the study physicians. This status will be assessed twice daily at 9AM and 5PM.
Patient experience | The patient's postoperative inpatient hospital stay, average 7 days
  In the patients who receive the AR game, responses to an electronic survey on the patient's experience designed by the MDACC Child Life team will be recorded when patients reach discharge-ready status.
Outpatient pain scores | 90 days after the patient is discharged from the hospital
  We will record average pain intensity experience by the patient during the 90-day (±10 Days) post surgery period. This data will be confirmed by direct contact to patient's guardian or as recorded in the electronic medical record during the patient's follow-up clinic visit
Outpatient quality of life | 90 days after the patient is discharged from the hospital
  Age-appropriate Pediatric Quality of Life Inventory (PedsQL) surveys will be administered to the patient (self-report) or guardian (proxy) by phone.

OTHER OUTCOMES:
Adverse events | Through study completion, average 4-month time period
  Any adverse events clinically determined to be related to the use of AR (i.e., falls) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Christina York, Principal Investigator — ALTality, Inc.; Juan Cata, MD, Principal Investigator — The University of Texas at Houston MD Anderson Cancer Center; Jamie Sinton, MD, Principal Investigator — The Texas Children's Hospital; Jae Eun Choi, Study Director — ALTality, Inc.
Locations (2):
- United States (2):
  - M.D. Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical data and statistical analyses included as a part of a publication will be shared with the scientific community per journal guidelines.